CLINICAL TRIAL: NCT00826020
Title: Prospective Evaluation of a Parenteral Omega-3 Fatty Acid Preparation (Omegaven™) in Therapy of Patients With TPN-Induced Cholestasis
Brief Title: Evaluation of Omegaven™ Parenteral Nutrition in Patients With Total Parenteral Nutrition (TPN)-Induced Cholestasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0084-09-FB
Record Dates: First submitted 2009-01-15; First posted 2009-01-21 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Parenteral Nutrition Associated Liver Disease PNALD; Cholestasis
Keywords: PN; parenteral nutrition; fat emulsions; omega-6 fatty acid; liver disease; fatty acid deficiency
MeSH Terms: conditions — Cholestasis; Hyperphagia; Liver Diseases | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omegaven™ (Experimental): This study will be a prospective, non-randomized, open-label study of Omegaven™ for provision of parenteral lipid calories. The study cohort, receiving the parenteral nutrition (PN) lipid at 1g/kg/day, will be compared to historical controls at University of Nebraska Medical Center (UNMC) where parenteral lipid calories were provided exclusively through soybean-based formulations. The study is planned to enroll 100 patients. The Intestinal Rehabilitation Program at UNMC sees between 20 and 30 new pediatric patients per year, with almost all being PN-dependent and over 75% presenting with a bilirubin ≥ 2mg/dL. Based on these calculations, we estimate 4-5 years to enroll 100 patients.
  Interventions: Drug: Omegaven™

INTERVENTIONS:
Drug: Omegaven™ — 10% Omegaven™, 50 or 100 mL bottle; 1gram/kg/day and is infused over 12-24 hours.
  Other Names: Omega-3 fat emulsion

SUMMARY:
The purpose of this study is to determine if established parenteral nutrition (PN) associated liver disease can be reversed or its progression halted by using a parenteral fat emulsion prepared from fish oil as measured by normalization of serum levels of hepatic enzymes and bilirubin.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the need for and time to small bowel transplantation or liver transplantation. This will be calculated as both the age at time of primary transplant as well as the length of time from initial evaluation to transplant.Secondary objectives are to determine if there are improvements in clinical measures associated with established parenteral nutrition- associated liver disease (PNALD). These will be determined by measurement of total and direct bilirubin levels, platelet count, serum albumin, and changes in both length and weight growth curves.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled in the Intestinal Rehabilitation Program at the University of Nebraska Medical Center, AND:
* Be unable to meet nutritional needs solely by enteral nutrition and be expected to require PN for at least another 30 days
* Have clinical evidence of parenteral nutrition associated liver disease (PNALD) as defined as a direct bilirubin of 2 mg/dl or more. A liver biopsy is desirable but not necessary for treatment
* Signed patient informed consent

Exclusion Criteria:

* Parent or guardian or child unwilling to provide consent or assent
* Inability or unwillingness on the part of parent/guardian or child to follow clinical recommendations of the Intestinal Rehabilitation Program
* Allergies or clinical conditions precluding safe use of Omegaven™

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Mercer, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Alwayn IP, Gura K, Nose V, Zausche B, Javid P, Garza J, Verbesey J, Voss S, Ollero M, Andersson C, Bistrian B, Folkman J, Puder M. Omega-3 fatty acid supplementation prevents hepatic steatosis in a murine model of nonalcoholic fatty liver disease. Pediatr Res. 2005 Mar;57(3):445-52. doi: 10.1203/01.PDR.0000153672.43030.75. Epub 2005 Jan 19. PMID 15659701
- [Background] Van Aerde JE, Duerksen DR, Gramlich L, Meddings JB, Chan G, Thomson AB, Clandinin MT. Intravenous fish oil emulsion attenuates total parenteral nutrition-induced cholestasis in newborn piglets. Pediatr Res. 1999 Feb;45(2):202-8. doi: 10.1203/00006450-199902000-00008. PMID 10022591
- [Background] Gura KM, Parsons SK, Bechard LJ, Henderson T, Dorsey M, Phipatanakul W, Duggan C, Puder M, Lenders C. Use of a fish oil-based lipid emulsion to treat essential fatty acid deficiency in a soy allergic patient receiving parenteral nutrition. Clin Nutr. 2005 Oct;24(5):839-47. doi: 10.1016/j.clnu.2005.05.020. PMID 16029913
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Diamond IR, Sterescu A, Pencharz PB, Kim JH, Wales PW. Changing the paradigm: omegaven for the treatment of liver failure in pediatric short bowel syndrome. J Pediatr Gastroenterol Nutr. 2009 Feb;48(2):209-15. doi: 10.1097/MPG.0b013e318182c8f6. PMID 19179884
- [Derived] Mercer DF, Hobson BD, Fischer RT, Talmon GA, Perry DA, Gerhardt BK, Grant WJ, Botha JF, Langnas AN, Quiros-Tejeira RE. Hepatic fibrosis persists and progresses despite biochemical improvement in children treated with intravenous fish oil emulsion. J Pediatr Gastroenterol Nutr. 2013 Apr;56(4):364-9. doi: 10.1097/MPG.0b013e31827e208c. PMID 23201707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment began May 1, 2008. The study was closed October 6, 2017
Groups:
- Omegaven™: This study will be a prospective, non-randomized, open-label study of Omegaven™ for provision of parenteral lipid calories. The study cohort, receiving the PN lipid at 1g/kg/day, will be compared to historical controls at UNMC where parenteral lipid calories were provided exclusively through soybean-based formulations. The study is planned to enroll 100 patients. The Intestinal Rehabilitation Program at UNMC sees between 20 and 30 new pediatric patients per year, with almost all being PN-dependent and over 75% presenting with a bilirubin ≥ 2mg/dL. Based on these calculations, we estimate 4-5 years to enroll 100 patients.
  Omegaven™: 10% Omegaven™, 50 or 100 mL bottle; 1gram/kg/day and is infused over 12-24 hours.
Period: Overall Study
Arm/Group | Omegaven™
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omegaven™
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: months] — Age at treatment start
  months | 5.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Gestational Age (weeks) [Mean (Standard Deviation); unit: weeks] | 31 (5)
Weight (kg) at Treatment Start [Mean (Standard Deviation); unit: kg] | 4.61 (2.09)
Weight Z Score at Treatment Start [Mean (Standard Deviation); unit: z-score] — The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean
  z-score | -1.60 (1.91)
Length (cm) at Treatment Start [Mean (Standard Deviation); unit: cm] | 55 (10)
Length Z Score at Treatment Start [Mean (Standard Deviation); unit: z score] — The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean
  z score | -2.09 (2.17)
Total Bilirubin (mg/dL) at Treatment Start [Mean (Standard Deviation); unit: mg/dL] | 9.9 (6.2)
Direct Bilirubin (mg/dL) at Treatment Start [Mean (Standard Deviation); unit: mg/dL] | 6.2 (3.9)
Serum aspartate aminotransferase (AST) at Treatment Start [Mean (Standard Deviation); unit: U/L] | 187 (137)
Serum alanine aminotransferase (ALT) at treatment Start [Mean (Standard Deviation); unit: U/L] | 159 (125)
Alkaline Phosphatase at Treatment Start [Mean (Standard Deviation); unit: U/L] | 436 (226)
Parenteral Nutrition (PN) Calories at Treatment Start (kCal/kg/d) [Mean (Standard Deviation); unit: kCal/kg/d] | 91 (11)
Enteral Calories at Treatment Start (kCal/kg/d) [Mean (Standard Deviation); unit: kCal/kg/d] | 8 (12)
Underlying Diagnosis [Count of Participants; unit: Participants]
  Necrotizing enterocolitis | 31
  Intestinal Atresia | 8
  Gastroschisis | 22
  Volvulus | 5
  Microvillus inclusion disorder | 4
  Intestinal Aganglionosis | 1
  Mesenteric Ischemia | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Progression to Small Bowel Transplantation.
Description: Whether or not the subject had an intestine-containing transplant or not
Time Frame: Bi-weekly x4, then monthly until the completion of the study, for an overall average of 5.5 years follow-up for the cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven™
Number analyzed (Participants) | 72
Participants | 19

2. Secondary Outcome: Number of Subjects With Reversal of Biochemical Cholestasis
Description: Of patients starting with elevated total serum bilirubin, the number that progress to normalization of serum total bilirubin in routine bloodwork
Time Frame: weekly x 4, then bi-weekly x4, then monthly until the completion of the study, with an average follow-up of 5.5 years for the study cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven™
Number analyzed (Participants) | 72
Participants | 56

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the term of the study, from May 1, 2009 until closure October 6, 2017. Each patient was assessed for treatment related adverse events from the initiation of therapy with Omegaven until 4 weeks after completion of therapy. This time was variable for each subject based on treatment length, with an overall average of 27 weeks follow-up for the cohort
Arm/Group | Omegaven™
All-Cause Mortality (participants affected / at risk) | 7/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-03-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT00826020/Prot_SAP_000.pdf